CLINICAL TRIAL: NCT07178080
Title: Comparative Analysis of PIUR Imaging Technology for Volume Reduction Rate Measurement in Thyroid Nodule Ablations
Brief Title: Comparing a New 3D Technology Used to Measure Thyroid Nodule Volume to Standard Ultrasound
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sarasota Memorial Health Care System (Other)
Responsible Party: Principal Investigator, Ralph Tufano, Principal Investigator, Sarasota Memorial Health Care System
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 25-ONC-49
Record Dates: First submitted 2025-09-07; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Nodules; Thyroid Nodule
Keywords: thyroid nodules; benign thyroid nodule; benign thyroid nodules; thyroid ablation
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: This is a double-blinded prospective study with a crossover design. Patients will serve as their own controls and receive a 2D ultrasound followed by a 3D ultrasound using PIUR technology at baseline, 2 weeks, 1 month, 3 months, 6 months, and 12 months. For the traditional 2D ultrasound scan, the physician will perform and interpret the scan to calculate volume reduction rates, following the American Thyroid Association (ATA) Thyroid Nodule Guidelines, which is the current standard of care. The PIUR 3D ultrasound results will be blinded to the physician to avoid bias during follow-up appointments.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 3D ultrasound using PIUR tUS Infinity (Experimental): Both imaging methods will be used throughout the study, the traditional 2D ultrasound followed by the 3D ultrasound using PIUR tUS Infinity. Volume measurements from each imaging method will be compared to one another.
  Interventions: Device: PIUR tUS Infinity Ultrasound
- Traditional 2D (Other): Both imaging methods will be used throughout the study, the traditional 2D ultrasound followed by the 3D ultrasound using PIUR tUS Infinity. Volume measurements from each imaging method will be compared to one another.
  Interventions: Device: PIUR tUS Infinity Ultrasound

INTERVENTIONS:
Device: PIUR tUS Infinity Ultrasound — PIUR imaging technology, cleared by the U.S. Food and Drug Administration under 510(k) (K240036), is designed to provide advanced volumetric imaging capabilities to improve accuracy in assessing nodule size and volume reduction.

SUMMARY:
After thyroid ablation procedure, the volume of the thyroid nodule (s) needs to be measured to see how well the procedure worked. Currently, these volumes are measured using traditional 2D ultrasound imaging. However, this approach comes with limitations because of the information 2D images cannot gather and because of differences in these measurements between different doctors. A new ultrasound technology called PIUR 3D imaging offers a novel alternative approach. The system uses advanced technology to create 3D images and can generate automated volume estimates. The PIUR imaging system, PIUR tUS Infinity, has been cleared by the Food and Drug Administration (FDA) to aid in treatment decisions when used alongside traditional 2D ultrasound imaging.

The purpose of this study is to test how effective and consistent the PIUR imaging technology is compared to standard 2D ultrasound in measuring thyroid nodule volume.

DETAILED DESCRIPTION:
PIUR imaging technology, cleared by the U.S. Food and Drug Administration under 510(k) (K240036), is designed to provide advanced volumetric imaging capabilities to improve accuracy in assessing nodule size and volume reduction. This technology has been validated for clinical use and shown to be equivalent to conventional methods. Currently, PIUR is intended to complement the diagnostic process and should not be used as the sole basis for treatment decisions. Instead, it serves as an adjunct to standard 2D ultrasound imaging.⁸ These features make PIUR a potential candidate for post-ablation monitoring of thyroid nodules, where precision and reproducibility are critical.

This study aims to compare the volume reduction rates obtained using PIUR imaging against those calculated by an experienced clinician using traditional 2D ultrasound. The findings will help assess whether PIUR offers a more reliable, operator-independent method for evaluating treatment outcomes following thyroid nodule ablation.

ELIGIBILITY:
Inclusion Criteria:

* 22 years old or older
* Patient of Dr. Ralph Tufano's office
* Undergoing thyroid nodule ablation
* The patient or their LAR must be willing and able to provide informed consent

Exclusion Criteria:

* Under 22 years of age
* Unable to undergo follow-up imaging
* Pregnancy
* Patients may be excluded at the physician's discretion based on their clinical judgement and/or if the health or safety of the patient may be potentially impacted by participating in this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-09-08 (Estimated); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
Thyroid nodule volumetric measurements | Will occur at baseline, 2 weeks, 1 month, 3 months, 6 months, and 1 year
  Compare thyroid nodule volumetric measurement readings retrieved from the PIUR 3D ultrasound and the volume calculated from a 2D ultrasound among patients having a thyroid ablation
Comparison of variability between measurements | Will occur at baseline, 2 weeks, 1 month, 3 months, 6 months, and 1 year
  Compare the variability in the thyroid nodule volume measurements between the PIUR 3D ultrasound and the variability calculated from a 2D ultrasound among patients having a thyroid ablation
Post-ablation thyroid volume reduction rate comparison | 2 weeks, 1-, 3-, 6-, and 12 months.
  Evaluate post-ablation thyroid volume reduction rates at 2 weeks and 1-, 3-, 6-, and 12 months in patients undergoing thyroid ablation and receiving PIUR 3D ultrasounds as compared to standard 2D ultrasounds.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Tufano, MD, Principal Investigator — Sarasota Memorial Health Care Systems
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trimboli P, Castellana M, Sconfienza LM, Virili C, Pescatori LC, Cesareo R, Giorgino F, Negro R, Giovanella L, Mauri G. Efficacy of thermal ablation in benign non-functioning solid thyroid nodule: A systematic review and meta-analysis. Endocrine. 2020 Jan;67(1):35-43. doi: 10.1007/s12020-019-02019-3. Epub 2019 Jul 20. PMID 31327158
- [Background] Bernardi S, Stacul F, Zecchin M, Dobrinja C, Zanconati F, Fabris B. Radiofrequency ablation for benign thyroid nodules. J Endocrinol Invest. 2016 Sep;39(9):1003-13. doi: 10.1007/s40618-016-0469-x. Epub 2016 Apr 20. PMID 27098804
- [Background] Durante C, Grani G, Lamartina L, Filetti S, Mandel SJ, Cooper DS. The Diagnosis and Management of Thyroid Nodules: A Review. JAMA. 2018 Mar 6;319(9):914-924. doi: 10.1001/jama.2018.0898. PMID 29509871
- See also: U.S. Food and Drug Administration. 510(k) Summary for PIUR Imaging Technology — https://www.accessdata.fda.gov/cdrh_docs/pdf24/K240036.pdf